CLINICAL TRIAL: NCT03878381
Title: Investigating the Wrinkle Reduction Potential of a Novel Compounded Skin Care Cream
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Steven D Daveluy, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1902002047
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Skin Care

STUDY DESIGN:
Intervention Model Description: Patients will engage in a split face trial, where each participant uses the vehicle on one side of the face and active ingredient treatment cream on the other side
Who Masked: Participant, Care Provider, Investigator
Masking Description: Block randomization will be utilized to determine which side will be the treatment side.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Compounded Skin Care Cream (Experimental): One side of the face will be randomly chosen as the treatment side
  Interventions: Combination Product: Skin Care Cream
- Placebo (Placebo Comparator): The other side of the face will be randomly chosen as the control
  Interventions: Drug: Placebo

INTERVENTIONS:
Combination Product: Skin Care Cream — The skin care regimen we will be testing includes ingredients such Hyaluronic acid 1%, Vitamin E Acetate, Vitamin A Acetate, Co-enzyme Q 10, L-Arginine, L-glutamine, Phytonadione, Argireline Peptide solution, GABA, Vitamin C, glycolic acid, and Fenugreek.
  Arms: Compounded Skin Care Cream
Drug: Placebo — The placebo will be a formula with no active ingredients
  Arms: Placebo

SUMMARY:
In the realm of cosmetics, skin care accounts for a significant share accounting for 35.3% of the global market, creating a $121 billion industry. While many of the products claim to have unique, natural formulations that boost skin care, many products contain chemicals that are potentially damaging to skin. Such ingredients include preservatives, parabens, fragrances, and formaldehyde, which can cause skin irritation and inflammation. Although these ingredients help to preserve the stability and longevity of products, it is plausible to achieve efficacy and improve skin structure without risking unnecessary damage.

The condition and health of the dermis rely largely on elastin, which gives the skin its elasticity, and collagen, which provides structure and strength. Collagen deteriorates naturally with age and exposure to environmental elements such as sunlight and toxins. Many skin rejuvenating interventions have focused on preventing the loss of collagen and elastin. The formulations used in this study will try to optimize cellular physiology, which in turn will create improvement in skin function, collagen strength, and wrinkle depth reduction. The skin care regimen we will be testing includes ingredients such Hyaluronic acid 1%, Vitamin E Acetate, Vitamin A Acetate, Co-enzyme Q 10, L-Arginine, L-glutamine, Phytonadione, Argireline Peptide solution, GABA, Vitamin C, glycolic acid, and Fenugreek. The chemicals used commercially have been avoided in this formulation to enhance the beneficial effects of the product.

The purpose of the study is to investigate the efficacy of a new skin care product utilizing the tools of complexion analysis software and optical coherence tomography(OCT). The primary endpoint will be a 15% reduction in facial wrinkles measured by complexion analysis software. Secondary endpoints will be a 10% reduction in skin roughness measured by OCT

DETAILED DESCRIPTION:
Patients will be advised to discontinue any other products, other than a mild cleanser, prior to beginning treatment. Patients will engage in a split face trial, where each participant uses the vehicle on one side of the face and active ingredient treatment cream on the other side. Baseline facial photography and OCT imaging will be performed on both sides of the face. One side of the face will be randomly chosen as the treatment side, and the other as an intrinsic control. Each day, the participant will wash their face in the morning with a standard cleanser, dry their face, then apply the medication to one side of their face and the vehicle to the other side of their face. The patient will then apply a standardized sunscreen SPF 30 to the entire face. Each night, the patient will again wash their face with the standard cleanser, and apply the two medications to the proper sides of the face. Patients will participate in a follow-up clinic visit 4 weeks, 8 weeks, 12 weeks and 16 weeks after beginning treatment. At each visit, photographs and OCT images will be taken of both sides of the face. At week 12, participants will take a survey to determine their satisfaction with the product and their subjective assessment of their skin changes and stop using the products and continue only the sunscreen. Four weeks after cessation of using the creams, they will return for photography and OCT imaging at a final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20 to 60

Exclusion Criteria:

1. Under age 20
2. Over age 60
3. Skin conditions such as rosacea, eczema, and allergic contact dermatitis limited to their face
4. Allergies to products being tested
5. Use of a facial anti-aging product within the past 6 weeks

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Reduction in Facial Wrinkle Count | 16 weeks
  The primary endpoint of this study is a 15% reduction in facial wrinkle count as measured by the Visia complexion analysis software.

SECONDARY OUTCOMES:
Reduction in Skin Roughness | 16 weeks
  A secondary endpoint of the study will be a 10% reduction in skin roughness as measured by an OCT image analysis

CONTACTS AND LOCATIONS:
Locations (1):
- WSUPG Dermatology, Dearborn, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halla N, Fernandes IP, Heleno SA, Costa P, Boucherit-Otmani Z, Boucherit K, Rodrigues AE, Ferreira ICFR, Barreiro MF. Cosmetics Preservation: A Review on Present Strategies. Molecules. 2018 Jun 28;23(7):1571. doi: 10.3390/molecules23071571. PMID 29958439
- [Background] Oba A, Edwards C. Relationships between changes in mechanical properties of the skin, wrinkling, and destruction of dermal collagen fiber bundles caused by photoaging. Skin Res Technol. 2006 Nov;12(4):283-8. doi: 10.1111/j.0909-752X.2006.00154.x. PMID 17026660
- [Background] Kulick MI, Gajjar NA. Analysis of histologic and clinical changes associated with Polaris WR treatment of facial wrinkles. Aesthet Surg J. 2007 Jan-Feb;27(1):32-46. doi: 10.1016/j.asj.2006.12.011. PMID 19341628
- [Background] Vasquez-Pinto LM, Maldonado EP, Raele MP, Amaral MM, de Freitas AZ. Optical coherence tomography applied to tests of skin care products in humans--a case study. Skin Res Technol. 2015 Feb;21(1):90-3. doi: 10.1111/srt.12161. Epub 2014 Jul 26. PMID 25066480
- [Background] Hibler BP, Qi Q, Rossi AM. Current state of imaging in dermatology. Semin Cutan Med Surg. 2016 Mar;35(1):2-8. doi: 10.12788/j.sder.2016.001. PMID 26963110